CLINICAL TRIAL: NCT07077694
Title: Accuracy of Artificial Intelligence Technology to Detect the Presence of Missed Canals of Endodontically Treated Mandibular Second Molar : Diagnostic Accuracy Experimental Study
Brief Title: Artificial Intelligence to Detect Missed Root Canals in Previously Treated Lower Back Teeth Using 3D Dental Imaging (CBCT)
Acronym: cone beam CT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Baheej Ghazi H Alhazmi, B.D.S, Future University in Egypt
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: FUE.REC(47)11-2024
Record Dates: First submitted 2025-07-01; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2024-10

CONDITIONS: Presence of Missed Canals; Morphological Variation
Keywords: Morphological variation; Presence of missed canals; CBCT; AI; Artificial intelligence; Clinical visual examination; dental operating microscope; mandibular second molar

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Presence of missed canals (Active Comparator)
  Interventions: Procedure: Root Canal Retreatment
- Morphological variation (Active Comparator)
  Interventions: Procedure: Root Canal Retreatment

INTERVENTIONS:
Procedure: Root Canal Retreatment — if Retreatment was needed, local anesthesia using 1.8 ml (one cartridge) of 4% articaine with 1:100,000 epinephrine local anesthetic solution, administered with end -loading cartridge aspirating syringe and a 27-gauge long needle. Under rubber dam isolation, All carious tissue and existing coronal restorations were thoroughly removed using a round bur, an endodontic access cavity, canal preparation and removal of existing root canal filling, irrigation with 2.6% NAOCL and saline, determining the working length using apex locator and PA radiograph, to be 0.5 to 1 mm shorter than radiographic apex, Drying the canal with paper point and obturation to achieve a dense, well adapted Monoblock obturation. A post-obturation periapical radiograph was taken to confirm the quality of the fill in terms of length, density, then sealed by a temporary restorative material.
  Other Names: Re-RCT

SUMMARY:
Aims to detect the Accuracy of Artificial Intelligence Technology in Detecting the Presence of Missed Canals of Endodontically Treated Mandibular Second Molar. Will Artificial intelligence software, CBCT and Clinical visual examination with dental operating microscope differs in the detection of presence of missed canals of endodontically treated human mandibular second molar ?

ELIGIBILITY:
Inclusion Criteria:

- 1) Patients must be medically free from any systemic disease that can affect root canal treatment.

2) Age range of the patient should be between 18 - 50 years old. 3) No sex predilection. 4) Patients must have good oral hygiene. 5) Patients with root canal-treated teeth. 6) Restorable teeth. 7) Positive patient acceptance for participating in the study. 8) Patients can sign informed consent.

Exclusion Criteria:

- 1) Patients with very poor oral hygiene. 2) Patients above 50 years and below 18 years. 3) Pregnant women after taking detailed history and pregnancy test must be in the first visit.

4) Psychologically disturbed patients. 5) Tooth periodontally affected with grade 2 or 3 mobility. 6) Non restorable teeth. 7) Tooth with abnormal anatomy and calcified canals.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-10-29 (Estimated); Study Completion 2025-10-29 (Estimated)

PRIMARY OUTCOMES:
Presence of missed canals | Pre Operative and At the end of the treatment within 1 week

SECONDARY OUTCOMES:
Morphological variation | Pre Operative and At the end of the treatment within 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine future university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided